CLINICAL TRIAL: NCT01338077
Title: A Multi-center, Double-blind, Randomized, Parallel Study to Evaluate the Efficacy and Safety of Sodium Alginate Oral Suspension (50 mg/ml) in Comparison to Omeprazole (20 mg/Cap) to Treat Non-erosive Gastro-esophageal Reflux Disease (NERD)
Brief Title: Efficacy and Safety of Sodium Alginate Oral Suspension to Treat Non-erosive Gastro-esophageal Reflux Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Cheng-Tang Chiu, Chief, Department of Gastroenterology and Hepatology, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TTYALG1001; CGMH-IRB-99-1495A3 (Other: ChangGungMH)
Record Dates: First submitted 2011-01-02; First posted 2011-04-19 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Gastroesophageal Reflux Disease; Heartburn
Keywords: Alginate; Gastroesophageal reflux disease
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Alginates; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sodium alginate (Experimental): Oral suspension, 50 mg/ml
  Interventions: Drug: Sodium alginate
- Omeprazole (Active Comparator): 20 mg/cap
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Sodium alginate — oral suspension, 50 mg/ml, 20 ml three times daily, 4 weeks
  Other Names: Alginos
  Arms: Sodium alginate
Drug: Omeprazole — 20 mg capsule, 1 capsule once daily, 4 weeks
  Other Names: Omelon
  Arms: Omeprazole

SUMMARY:
About 60% of patients with typical gastroesophageal reflux symptoms such as heartburn and regurgitation are considered to have non-erosive reflux disease (NERD). Patients with NERD show an overall poorer response to PPI treatment than patients with erosive reflux disease. Sodium alginate oral suspension is a medication indicated for the relief of gastroesophageal reflux symptoms. This multi-center, double blind, randomized trial aims to compare the efficacy and safety profiles of sodium alginate oral suspension (50 mg/ml) 20 ml three times daily with that of omeprazole (20 mg/capsule) 1 capsule once daily for the treatment of NERD patients in Taiwan. Efficacy assessments include percentage of patients achieving adequate relief of heartburn or regurgitation after 4 weeks treatment, improvement of reflux symptoms as assessed by reflux disease questionnaire before and after treatment, and patients overall satisfaction at the end of study. Safety assessments include incidence of adverse events and change of the laboratory test results. The study hypothesis is that treatment with sodium alginate is non-inferior to omeprazole in relieving heartburn or regurgitation symptoms of the NERD patients.

DETAILED DESCRIPTION:
This multi-center, double blind, randomized trial aims to compared the efficacy and safety profiles of sodium alginate oral suspension (50 mg/ml) 20 ml three times daily with that of omeprazole (20 mg/capsule) 1 capsule once daily for the treatment of non-erosive reflux disease (NERD) patients in Taiwan. Patients will be included into study if they are diagnosed as NERD; with heartburn or regurgitation (either one) as main symptom at least 2 days a week and had been present for ≧1 month before screening; with heartburn or regurgitation (either one) during the 7 days screening period, either with frequency for ≧4 days of mild symptom, or ≧ 2 days of moderate to severe symptom; and have signed the informed consent. Patients will be excluded if they are diagnosed as erosive gastroesophageal reflux disease (GERD), Barrett's esophagus or esophageal stricture; with active or healing gastroduodenal ulcer (except scars); with history of gastric, duodenal or esophageal surgery; with intrahepatic stone, gallstone, gallbladder sludge, hepatic or pancreatic carcinoma as evidenced by abdominal ultrasonography, with ischemic heart disease as evidenced by electrocardiogram; taking a proton pump inhibitor (PPI) within 14 days before screening, or a H2-blocker, prokinetic agent or antacid within 7 days before screening; or with clinically significant liver or kidney disease. The primary efficacy endpoint is percentage of patients achieving adequate heartburn (defined as a burning feeling or pain behind the breast bone) or regurgitation (defined as an acid taste in the mouth or unpleasant movement of material upwards from the stomach) relief at day 28 as assessed by patient diary. The secondary efficacy endpoints are percentage of patients achieving adequate heartburn or regurgitation relief at day 14; change from baseline of the reflux disease questionnaire total score at day 14 & 28; patients' overall satisfaction at the end of study; and number of antacid used during the 4-week treatment period. The safety endpoints are incidence of adverse events, and changes in laboratory test results (hematology, biochemistry, and urinalysis). The study hypothesis is that treatment with sodium alginate is non-inferior to omeprazole in relieving heartburn or regurgitation symptoms of the NERD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age of 20-75 years old (inclusive) in Taiwan of both genders
* Out-patients who had been diagnosed as non-erosive gastroesophageal reflux disease (NERD)
* Patients with heartburn or regurgitation (either one) as main symptom at least 2 days a week and had been present for > or = 1 month before screening
* Patients with heartburn or regurgitation (either one) during the 7 days screening period, either with frequency for > or = 4 days of mild symptom, or for > or = 2 days of moderate to severe symptom
* Patients have signed the informed consent form

Exclusion Criteria:

* Patients with erosive gastroesophageal reflux disease (GERD), Barrett's esophagus or esophageal stricture
* Patients with active or healing gastroduodenal ulcer (except scars)
* Patients with history of gastric, duodenal or esophageal surgery
* Patients with malignant disease of any kind
* Patients with intrahepatic stone, gallstone, gallbladder sludge, hepatic or pancreatic carcinoma as evidenced by abdominal ultrasonography
* Patients with ischemic heart disease as evidenced by electrocardiogram
* Female patients who are pregnant or nursing mother
* Patients with a history of allergy to any of the study drugs or their related compounds
* Patients with a history of alcohol or drug abuse
* Patients with clinically significant liver disease (aspartate aminotransferase (AST), alanine aminotransferase (ALT)>2 upper limits of normal)
* Patients with clinically significant renal disease (serum creatinine >1.5 mg/dl)
* Patients taken a proton pump inhibitor (PPI) within 14 days before screening, or a H2-blocker, prokinetic agent or antacid within 7 days before screening
* Patients participated any investigational drug trial within 4 weeks before screening
* Patients with any other conditions or diseases that investigator considers it is not appropriate to enter the study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients achieving adequate heartburn or regurgitation relief at day 28 as assessed by patient diary | 4 weeks
  Adequate heartburn or regurgitation relief is defined as no more than 1 day of mild heartburn or regurgitation episodes in the last 7 days before day 28

SECONDARY OUTCOMES:
Percentage of patients achieving adequate heartburn or regurgitation relief at day 14 as assessed by patient diar | 2 weeks
  Adequate heartburn or regurgitation relief is defined as no more than 1 day of mild heartburn or regurgitation episodes in the last 7 days before day 14
Change from baseline of the Reflux Disease Questionnaire (RDQ) total score at days 14 & 28 | 2 and 4 weeks
  RDQ is a 12-item self-administered questionnaire and there are 3 subscales that evaluate frequency and severity of heartburn, regurgitation and dyspepsia. Each item is scored on a 6-point Likert scale ranging from 0 to 5. The RDQ total scores are determined by the sum of 12-item scores.
Patients' overall satisfaction at the end of study | 4 weeks
  The overall satisfaction is categorized as:0=very poor; 1=poor; 2=unsatisfactory; 3=satisfactory; 4=good; 5=very good
Number of antacid used during the treatment period | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Tang Chiu, MD, Principal Investigator — Chief, Department of Gastroenterology and Hepatology, Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Chiu CT, Hsu CM, Wang CC, Chang JJ, Sung CM, Lin CJ, Chen LW, Su MY, Chen TH. Randomised clinical trial: sodium alginate oral suspension is non-inferior to omeprazole in the treatment of patients with non-erosive gastroesophageal disease. Aliment Pharmacol Ther. 2013 Nov;38(9):1054-64. doi: 10.1111/apt.12482. Epub 2013 Sep 11. PMID 24024757